CLINICAL TRIAL: NCT03987178
Title: Microbiologic Alterations of the Conjunctiva of Hot Tub-soaking Ophthalmologists
Acronym: MACHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-26141
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Conjunctivitis, Bacterial; Keratitis Bacterial
Keywords: hot tub; conjunctival cultures; bacterial keratitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — dunk protein, Drosophila

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: A provider is assigned to perform conjunctival swabs; this person is completely masked to exposure. The culture plates, which are randomized, are sent to a microbiology lab and the technicians are completely masked to exposures when reading the plates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head Dunk (Experimental): Subjects who are assigned to be in this arm are asked to sit in a hot tub for 15 minutes and instructed to submerge his or her head in the hot tub at least once and at least up to the eyebrows during his or her time in the hot tub.
  Interventions: Behavioral: Dunk; Other: Exposure to Hot Tub
- No Head Dunk (Placebo Comparator): Subjects assigned to this arm are asked to sit in a hot tub for 15 minutes but to keep his or her chin above water during the entire time.
  Interventions: Other: Exposure to Hot Tub

INTERVENTIONS:
Behavioral: Dunk — If randomized to "Dunk," the subject is asked to submerge his or her head in the hot tub at least up to brow level.
  Arms: Head Dunk
Other: Exposure to Hot Tub — Subjects will be asked to sit in a hot tub for 15 minutes (with an individual timer).

SUMMARY:
The purpose of this study is to determine if there are microbiologic alterations of the ocular surface after hot tub exposure. The study will evaluate the number of microbes before and after hot tub use in order to find out whether hot tub exposure has any change on the organisms present on the ocular surface. Participants will be randomized to dunk or not to dunk their head during their time in the hot tub.

DETAILED DESCRIPTION:
Keratitis is a rare destructive cause of blindness. It typically affects young and healthy individuals, is excruciatingly painful, and difficult to treat. With 60% of cases mis-diagnosed at presentation, acanthamoeba keratitis carries a far worse visual prognosis compared to other cornea infections. Exposure to hot tubs is a widely accepted risk factor. However, the mechanism of infection and prediction of who is at risk is unknown as the vast majority of hot tub users do not become infected.In vivo changes to ocular microbiology after hot tub exposure has never been described.

Changes to ocular microbiology after exposure to hot tubs have not been described. The purpose of this study is to investigate whether there are significant alterations in the microbiology of the conjunctiva after hot tub exposure that may contribute to these changes.

This study will recruit at least 34 subjects, who will be randomized to head submersion versus no head submersion, using at least three different hot tubs. A conjunctival swab, a minimal-risk test performed routinely in the eye clinic, will be performed before and after 15 minutes of hot tub exposure on one eye (randomized) per subject. The swabs will be plated on blood agar (bacterial cultures) and non-nutrient agar (acanthamoeba cultures).

In this prospective study, healthy subjects will be recruited. The study will be Health Insurance Portability and Accountability Act compliant and approved by the Institutional Review Board. All subjects will review and sign an informed consent form.

Each patient will have the conjunctiva of one eye (randomized) cultured. This practically no-risk technique entails touching a polyester-tip swab to the lining of the lower eyelid. Each subject will be randomized to head submersion or no head submersion; this exposure will be masked by the study coordinator. After 15 minutes of hot tub exposure, the subject will have the same eye swabbed for cultures.

Each sample (pre- and post-hot tub) will be randomly assigned a study number. One study coordinator will record and mask data. Water from each tub will be cultured.

The culture plates will be sent to our microbiology facility at UCSF and identification of organisms on the blood agar plates will be performed on our MALDI (mass spectrometry to identify bacteria and fungi). Non-nutrient agar plates will be plated with E. coli overlay and incubated for up to 7 days. The plates will be randomized and the microbiologists will be masked to exposures.

ELIGIBILITY:
Inclusion criteria:

* greater of 18 years of age
* a willing participant
* healthy

Exclusion criteria:

* pregnancy
* high or low blood pressure
* active diarrhea
* lymphedema
* heart disease
* seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Quantity of organisms | 1 year
  Genus-species will be identified for each sample, and quantified with an ordinal scale (0-4). The total of this score will be the quantity for that person-time. The primary analyses will be a Wilcoxon Rank Sum test (Mann-Whitney) between the two arms at the follow-up time point (randomized comparison of dunk vs no-dunk), and a Wilcoxon Signed Rank test between pre-hot-tub and post-hot-tub (longitudinal comparison of all cases).
  We estimate that a total of 20 subjects will provide 80% power to detect a 1.25 SD difference in the total quantity score between randomization arms at the post (f/u) time point. We estimate 80% power to detect a .9 SD difference between pre (baseline) and post (f/u) time points in a paired longitudinal analysis.

SECONDARY OUTCOMES:
Richness (number of species per sample) of organisms found in the conjunctiva with hot tub use (post-test comparison) | 1 year
  The investigators will assess whether organism diversity (richness) changes between arms (post-test comparison) using Simpson's Diversity, expressed in units of effective number (see Jost). We will also assess using Shannon's Diversity.
Richness (number of species per sample) of organisms found in the conjunctiva with hot tub use (pre versus post) | 1 year
  The investigators will assess whether organism diversity (richness) changes longitudinally (pre vs post-test comparison).
Difference in organism profile with hot tub use (pre versus post) | 1 year
  The investigators will determine whether the organism profile differs longitudinally (pre vs post-test comparison) using L-2 norm (Euclidean distance) and PERMANOVA. We will also assess using L-1 norm (Manhattan distance)
Difference in organism profile with hot tub use (between arms) | 1 year
  The investigators will determine whether the organism profile differs between arms (post-test comparison) using L-2 norm (Euclidean distance) and PERMANOVA. We will also assess using L-1 norm (Manhattan distance)
Quantity comparing pre-hot tub and post-hot tub swabs | 1 year
  We will compare quantity of organisms (amount and type) before and after hot tub use in both arms. We will used a paired t-test for analysis.
Specific organisms found in the conjunctiva with hot tub use | 1 year
  The investigators will compare specific organisms (Staphylococcus epidermidis, Corynebacterium species) between arms (post-test only) and longitudinally between time points (pre vs post-test) with Bonferroni correction

CONTACTS AND LOCATIONS:
Overall Officials: Gerami D Seitzman, MD, Principal Investigator — UCSF/Proctor Foundation
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No